CLINICAL TRIAL: NCT00391495
Title: Inflammation in Children With Attention-Deficit/Hyperactivity Disorder
Acronym: ADHD_CYTO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TASMC-06-NV-246-CTIL
Record Dates: First submitted 2006-10-22; First posted 2006-10-24 (Estimated); Last update posted 2007-06-19 (Estimated); Status verified 2006-08

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD; Cytokines; CR-P
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Blood drawing

SUMMARY:
The aim of this study is to investigate the inflammatory response in children with this disorder.

DETAILED DESCRIPTION:
Attention deficit-hyperactivity disorder (ADHD) is a prevalent childhood neuropsychiatric disorder, characterized by age-inappropriate and impairing levels of inattention, hyperactivity and impulsiveness. Approximately 5-10% of school-age children are affected by ADHD, and in many cases, symptoms persist into adolescence and adulthood.

Cytokines are key mediators of immune function and can be either pro-inflammatory or anti-inflammatory. Recently few studies have suggested involvement of cytokine pathways in subjects with ADHD.

Polymorphism of IL-1 receptors antagonists' alleles have been suggested in families and subjects suffering from ADHD. Moreover, a new variant of inflammatory bowel disease, another immunological based disease, was recently suggested in children with ADHD and other developmental disorders. There are no other published reports on cytokine production in children who suffer from ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. A defined condition of ADHD according to TOVA test (TOVA score > (-1.8), Connor's questionnaire (Connor's score > 15 points) and Achenbach's questionnaire;
2. A consent form signed by parents or legal guardianships;

Exclusion Criteria:

1. A history of any other neurological or major psychiatric disorder or other significant medical problems;
2. No current medications;

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2007-09; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Prof. (MD), Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- The Unit of Clinical Nutrition, Tel Aviv, Israel